CLINICAL TRIAL: NCT06587399
Title: Comparison of Manual Therapy Versus Low-medium Energy Radial Shock Waves in the Treatment of Subacromial Syndrome in a Randomized Clinical Trial
Brief Title: Comparison of Manual Therapy Versus Radial Shock Waves in the Shoulder Pain Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/2024/3/053
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Impingement; Shoulder Pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy treatment (Active Comparator): Joint mobilization techniques in the shoulder together with the treatment of muscle trigger points using pressure release techniques
  Interventions: Other: Manual therapy treatment
- Radial shock wave treatment (Experimental): Low-medium energy radial shock waves will be used to treat muscle trigger points and the insertion of the supraspinatus muscle
  Interventions: Other: Radial shock wave treatment

INTERVENTIONS:
Other: Manual therapy treatment — Joint mobilization techniques will be applied to the shoulder joint complex, adapted to the subjects' degree of irritability.
  The muscular trigger points of the shoulder muscles will be treated using a pressure release technique applied for 60 seconds.
  In addition, the subjects will carry out a 12-week home-based therapeutic exercise program.
  Arms: Manual therapy treatment
Other: Radial shock wave treatment — The treatment will be carried out with 1 session per week for 6 weeks. For this purpose, a radial shock wave generator will be used, at a frequency of 8 to 12 Hz, 2000 pulses/session and with a pressure of 2.5 to 4.0 bar.
  Between 3 and 5 points will be treated per session: insertion of the supraspinatus muscle, dorsolateral area under the acromion and a maximum of 3 trigger points of the rotator cuff muscles.
  In addition, the subjects will carry out a 12-week home therapeutic exercise program.
  Arms: Radial shock wave treatment

SUMMARY:
Subacromial syndrome represents the third leading cause of pain in the general population. There is no clear pathophysiological explanation, nor a specific treatment. Manual therapy stands out as one of the reference treatments for this disease, however, it is complex to develop a specific protocol. On the other hand, shock waves have still not received adequate attention in the treatment of this pathology. The aim of this study will focus on using manual treatment using ischemic pressure, joint mobilizations and myofascial techniques in comparison to shock wave therapy to determine which is more effective.

This study will be a randomized, single-blind clinical trial with third-party evaluation. In it 88 subjects suffering from subacromial syndrome will participate. 44 patients will receive treatment through manual therapy over 6 weeks and other 44 patients through low-med energy radial shock waves for 6 weeks.

All subjects will complete their treatment with a 12-week home-based therapeutic exercise program.

The main endpoint of the study will be pain measured using the visual analogue scale (VAS) in motion. Pain will also be assessed using the VAS scale at rest and overnight. The Spadi Spanish version questionnaire will be used, shoulder strength will be measured using a handheld dynamometer and the ranges of motion will be measured.

Data will be measured before and one year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral shoulder pain with no history of trauma.
* Pain of at least 4/10 on the Visual Analogue Scale for a minimum period of 3 months.
* Be positive in at least 3 of the following 5 tests: painful arc test, Neer impingement test, Hawkins-Kennedy test, Jobe test, external rotation test against resistance for the infraspinatus tendon.

Exclusion Criteria:

* Presence of red flags.
* Diagnosis of shoulder instability.
* Diagnosis of frozen shoulder.
* Diagnosis of complete rupture of the common rotator cuff tendon.
* Diagnosis of cervical radiculopathy.
* Diagnosis of whiplash.
* Diagnosis of degenerative disease of the glenohumeral joint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | Change from Baseline pain at 12 month.
  Pain intensity will be measured using the Visual Analog Scale (VAS) for pain. The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and ten the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.

SECONDARY OUTCOMES:
Disability | Change from Baseline pain at 12 month.
  Disability will be measured by Shoulder Pain and Disability Index (SPADI).The Spanish version of SPADI has high test-retest reliability (ICC 0.89-0.93).The clinically important minimum difference varies between 8 and 13.2. The minimum value is 0 and de maximum value is 100
Muscle Force | Change from Baseline pain at 12 month.
  Force will be measured by a manual dynamometer (microFET®2, Hoggan Scientific LLC). Measurements will be taken in Newtons (N). It will be evaluated in the movements of external rotation and abduction of both shoulders.
  Manual dynamometry has proven to be a tool with excellent intra-examiner reliability to assess isometric force in external rotation of the shoulder, with an intraclass correlation coefficient (ICC) of 0.96 (0.93-0.98). The minimum value is 0 and de Maximum values is 55
Graded Chronic Pain Scale (CPGS) | Change from Baseline pain at 12 month.
  The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. It is suitable for use in all chronic pain conditions.The 3 subscale scores (characteristic pain intensity, disability score, and the disability points score) are used to classify subjects into 1 of the 5 pain severity grades: grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting.
Shoulder range of movement (ROM) | Change from Baseline pain at 12 month.
  Active range of motion of glenohumeral joint will be measured using a Standard BASELINE ® 12-inch plastic goniometer following previous guidelines. The 0 degrees of movement is worse and 180 degrees is the better

CONTACTS AND LOCATIONS:
Locations (1):
- Alcalá University, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No